CLINICAL TRIAL: NCT04409236
Title: Randomized Trial of a Smartphone Application to Help Cancer Patients Stop Smoking (Quit2Heal)
Brief Title: Quit2Heal Smartphone App in Helping Cancer Patients Quit Smoking
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); American Cancer Society, Inc. (Other); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RG1007577; NCI-2020-03442 (Other Grant/Funding Number: CTRP (Clinical Trial Reporting Program)); 10432 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA253975 (NIH)
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Quit2Heal app) (Experimental): Patients receive the Quit2Heal app and are encouraged to use it frequently. During the entire 12-month follow-up period, the app will remain fully available anytime study participants wish to use it.
  Interventions: Behavioral: Quit2Heal; Other: Survey Administration
- Arm II (QuitGuide app) (Active Comparator): Patients receive the QuitGuide app and are encouraged to use it frequently. During the entire 12-month follow-up period, the app will remain fully available anytime study participants wish to use it.
  Interventions: Behavioral: QuitGuide; Other: Survey Administration

INTERVENTIONS:
Behavioral: Quit2Heal — Use Quit2Heal app
  Other Names: Quit2Heal App; Quit2Heal Smartphone App; Quit2Heal Smartphone Application
  Arms: Arm I (Quit2Heal app)
Behavioral: QuitGuide — Use QuitGuide app
  Other Names: QuitGuide App; QuitGuide Smartphone App; QuitGuide Smartphone Application
  Arms: Arm II (QuitGuide app)
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase III trial compares the Quit2Heal smoking cessation smartphone application (app) to the QuitGuide app in helping cancer patients quit smoking. Both apps provide tools to cope with urges to smoke, step-by-step guides for quitting smoking, help in planning for quitting and staying tobacco-free, and scientifically-based recommendations for how to select medications that aid in smoking cessation.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive the Quit2Heal app and are encouraged to use it frequently. During the entire 12-month follow-up period, the app will remain fully available anytime study participants wish to use it.

ARM II: Patients receive the QuitGuide app and are encouraged to use it frequently. During the entire 12-month follow-up period, the app will remain fully available anytime study participants wish to use it.

After randomization, patients are followed up at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosed with cancer within the past 24 months or currently receiving or planning to receive cancer treatment in the next 3 months
* Smoked a cigarette (even a puff) in the past 30 days
* Interested in learning skills to quit smoking
* Willing to be randomly assigned to either smartphone application
* Live in the United States and will remain in the United States (US) for the next 12 months
* Have at least daily access to their own smartphone
* Know how to download a smartphone application
* Be willing and able to read English
* Not currently (i.e., within past 30 days) using other smoking cessation interventions
* Have never participated in our prior research trials
* Have never used the National Cancer Institute (NCI)'s QuitGuide app
* Being willing to complete a follow-up survey at 3, 6, and 12 months post-randomization
* Providing email, phone number(s), and mailing address

Exclusion Criteria:

* Currently (i.e., within past 30 days) using other smoking cessation interventions
* Has participated in our prior research trials
* Has used the NCI's QuitGuide app
* Not willing to complete a follow-up survey at 3, 6, and 12 months post-randomization
* Not providing email, phone number(s), and mailing address

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2026-09-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with 30-day cigarette smoking cessation at 12 months. | At 12 months after randomization
  No smoking at all in the past 30 or more days.

SECONDARY OUTCOMES:
Number of participants with 30-day cigarette smoking cessation at 3 months. | At 3 months after randomization
  No smoking at all in the past 30 or more days.
Number of participants with 30-day cigarette smoking cessation at 6 months. | At 6 months after randomization
  No smoking at all in the past 30 or more days.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Bricker, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT04409236/ICF_000.pdf